CLINICAL TRIAL: NCT04553822
Title: Effectiveness of Mucociliary Clearance Techniques in Non-hospitalized Moderate Bronchiolitis: a Multicenter Clinical Trial
Brief Title: Mucociliary Clearance Techniques in Moderate Bronchiolitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guadarrama Hospital (Other)
Collaborators: Fisiobronquial Clínicas (Other)
Responsible Party: Principal Investigator, J. Nicolas Cuenca Zaldivar, Rehabilitation Service Principal Investigator, Guadarrama Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 9.0
Record Dates: First submitted 2020-09-12; First posted 2020-09-17 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Bronchiolitis
Keywords: Physical Therapy; Respiratory; Pediatric
MeSH Terms: conditions — Bronchiolitis | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Single-blind randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Single (Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Assisted autogenous drainage group (DAA) (Experimental): The technique consists of positioning the patient in a supine position with the head slightly elevated on the supporting plane and then placing both hands around the rib cage and applying bimanual expiratory compression on both hemithoraxes.
  Interventions: Other: Assisted autogenous drainage group (DAA)
- Group prolonged slow expiration (ELPr) (Experimental): This technique is applied to the baby by means of a slow thoracic-abdominal pressure that begins at the end of a spontaneous expiration and continues until the residual volume.
  Interventions: Other: Group prolonged slow expiration (ELPr)
- Control group (CG) (Active Comparator): Nebulization with 4 ml Muconeb® 3% hypertonic serum, for 8 minutes in a Philips® vibrating mesh nebulizer.
  Interventions: Other: Control group (CG)

INTERVENTIONS:
Other: Assisted autogenous drainage group (DAA) — DAA, is used when the patient is not able to perform this technique autonomously and is assisted by the physiotherapist. Its greatest utility is in infants and preschoolers. The technique consists of positioning the patient in a supine position with the head slightly elevated on the supporting plane and then placing both hands around the rib cage and applying bimanual expiratory compression on both hemithoraxes. The physiotherapist must ensure that the child takes 2 to 3 controlled breaths, close to the residual level, with the objective that the expiratory flow displaces the secretions, located distally, towards the central airways.
  Arms: Assisted autogenous drainage group (DAA)
Other: Group prolonged slow expiration (ELPr) — Passive expiratory aid technique applied to the baby by means of a slow thoracic-abdominal pressure that begins at the end of a spontaneous expiration and continues until the residual volume. The physiotherapist through the provoked cough or stimulation of the trachea achieves the expectoration of the sputum.
  Arms: Group prolonged slow expiration (ELPr)
Other: Control group (CG) — Nebulization with 4 ml Muconeb® 3% hypertonic serum, for 8 minutes in a Philips® vibrating mesh nebulizer. Once the nebulization is finished, you will wait 30 minutes in a closed room.
  Arms: Control group (CG)

SUMMARY:
Acute viral bronchiolitis (BE) is an inflammatory disease of the lower respiratory tract, with a viral etiology, where the respiratory syncytial virus is the most prevalent agent. Respiratory physiotherapy (FTR) aims to remove airway obstruction, which decreases airway resistance, improves gas exchange, and reduces respiratory load. It is widely used in the treatment of children with chronic respiratory disease, but has long been debated as a treatment for bronchiolitis.

The objective of this study is to evaluate the effectiveness of two mucociliary clearance techniques in non-hospitalized children <12 months with a first episode of moderate BE.

This is a clinical trial that aims to recruit patients from 2 to 12 months who attend the Physiobronchial physiotherapy centers in Madrid, A Coruña, and Barcelona with a first-time medical diagnosis of BQ of 48 hours of maximum evolution. Participants will be randomly assigned into 3 groups: Group A: Assisted Autogenous Drainage (DAA), Group B: Prolonged Slow Expiration (ELPr) and Control Group. The main variables are the Acute Bronchiolitis Severity Scale (ESBA), oxygen saturation (SaO2), the modified Wood-Downes scale (WD-S), the Hospital scale Sant Joan de Déu (HSJD) and the ReSVinet Scale (RSV-S), and will be measured by a blinded evaluator at the beginning of the session (T0), 20 minutes after administering short-acting β2 adrenergic agonist (SABA) (T20 ), immediately after nebulization (T40) and at the end of the physiotherapist's intervention (T60). It will be reassessed 48 hours after the session (T48h) and the protocol will be repeated completely if it has not dropped at least two points according to the scales.

DETAILED DESCRIPTION:
The main objective of the present work is to evaluate the effectiveness of two mucociliary clearance techniques in non-hospitalized children <12 months with a first episode of moderate BE.

Once each patient legal guardians has signed the informed consent document and it has been verified that the inclusion criteria are met, participants will be assigned the same identification number (ID) that is related to its Clinical History (CH) by simple coding; custody of the file with the relationship of each ID with its CH will be the responsibility of the principal investigator. The method of blinding in the allocation will be performed by choosing opaque sealed envelopes by a person external to the study. The contents of the envelopes will be the random assignment cards to each of the three groups, this simple random numerical sequence will be generated by computer using the R program see 3.5.1. (R Foundation for Statistical Computing,Institute for Statistics and Mathematics, Welthandelsplatz 1, 1020 Vienna, Austria) based on stratified sampling for homogeneity, in three groups:Group A: assisted autogenous drainage group (DAA), group B: group prolonged slow expiration (ELPr), group C: control group (CG).

None of the children that make up both intervention group A and B, and the control group, will be prohibited from the usual pharmacological treatment prescribed by their doctor. It will collect in the investigator's notebook the medications that each patient has prescribed by their doctor. Physiotherapists cannot prescribe drugs, but can administer them at the beginning of the protocol after the prescription by the doctor.

Within the protocol, the short-acting β2 adrenergic agonist (SABA) will be administered, prior to nebulization with 4 ml Muconeb® 3% hypertonic serum, for 8 minutes in a Philips® vibrating mesh nebulizer. Next, following protocols will be applied:

* Intervention based on DAA Group A: the technique consists of positioning the patient in a supine position with the head slightly elevated on the supporting plane and then placing both hands around the rib cage and applying bimanual expiratory compression on both hemithoraxes. The physiotherapist must ensure that the child takes 2 to 3 controlled breaths, close to the residual level, with the objective that the expiratory flow displaces the secretions, located distally, towards the central airways.
* Intervention based on ELPr Group B: this technique applied to the baby by means of a slow thoracic-abdominal pressure that begins at the end of a spontaneous expiration and continues until the residual volume. The physiotherapist through the provoked cough or stimulation of the trachea achieves the expectoration of the sputum.
* Group C: nebulization with 4 ml Muconeb® 3% hypertonic serum, for 8 minutes in a Philips® vibrating mesh nebulizer.

The timing of intervention protocol will be followed: a) The SABA prescribed by the doctor will be administered to all patients; b) 20 minutes later the patient will then receive an 8-minute nebulization of Muconeb® 3% hypertonic solution; c) The treatment techniques protocol will consist of a standard 20 minute session based on nasal washes and the protocols descrive above for each intervention group.

Both groups will receive 3 evaluations by an investigator who will be blinded on the treatment and the objectives. The evaluations will be carried out at the beginning of the session (T0), 20 minutes after the SABA administration (T20), after the nebulization of Muconeb® 3% hypertonic solution (T30), after intervention treatment protocol (T60) and, finially, after 48 hours from ending treatment session (T48).

The main variables will classify the participants according to the initial clinical severity score proposed by the Acute Bronchiolitis Severity Scale (ESBA), the Wood-Downes Scale modified by Ferres (WDF-S), the Scale of the Sant Joan de Déu Hospital (HSJD) and the ReSVinet Scale (RSV-S). HR is a variable that is collected on the HSJD and WDS scales. SaO2 is included in the HSJD and ESBA scale, both will be measured through a pulse oximeter (Radical Touchscreen from Massimo®, Masimo Corporation, Irvine, CA).

ELIGIBILITY:
Inclusion Criteria:

* Be between 2 and 12 months of age (according to the latest Clinical Practice Guide on BQ of the National Health System available in Spain, it is considered comorbidity to have less than 2 months old)twenty.
* Have a medical diagnosis of a first episode of acute BE.
* Acute BE with a moderate degree of involvement with a score on the Acute Bronchiolitis Severity Scale (ESBA) ≥ 5 and ≤ 9.
* Acute BE with a degree of moderate severity with a modified Wood-Downes Scale (WD-S) score ≥ 4 and ≤ 5.
* Acute BE in a moderate degree of severity with a score according to the Hospital Sant Joan de Déu (HSJD) scale ≥ 6 and ≤ 10.
* Acute BE in a moderate degree of severity with a score on the ReSVinet Scale ( RSV-S) ≥ 7 and ≤ 13.
* Have not previously received respiratory physiotherapy since diagnosis.
* Oxygen saturation (SaO2) ≥ 94%,and j) have the informed consent of the child's legal guardians.

Exclusion Criteria:

* Acute BE with a score of ≤ 4 or ≥ 10 according to ESBA.
* Acute BE with a score ≤ 3 or ≥ 6 on the WD-S.
* Acute BE with score ≤ 5 or ≥ 11 in HSJD.
* Acute BE with score ≤ 6 or ≥ 14 in RSV-S, f) SaO2 ≤ 93%.
* Associated congenital heart disease, h ) previous hospitalizations for recurrent wheezing or episode of bronchiolitis requiring admission for more than 48 hours.
* Medical diagnosis of recurrent wheezing.
* Failure to follow up at 48 hours.
* No parental consent.
* Premature infants <32- 35 weeks.
* Bronchopulmonary dysplasia.

Ages: 2 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 165 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-03-06 (Actual); Study Completion 2022-04-06 (Actual)

PRIMARY OUTCOMES:
Acute Bronchiolitis Severity Scale | 48 hours
  Is a quantitative cumulative scale designed to assess clinical severity in patients with BE. The clinical severity scoring system is made up of five items: wheezing or crackles (only the one with the highest score is taken into account), effort, i / e ratio, RR and HR. Each item is scored from 0 to 4, the values of each item are added and a total result of (0-4) mild, (5-9) moderate and (10-13) severe is obtained, with 13 being the maximum score and 0 the minimum.

SECONDARY OUTCOMES:
Wood-Downes Scale modified by Ferres (WDF-S) | 48 hours
Scale of the Sant Joan de Déu Hospital | 48 hours
  Is a quantitative cumulative scale designed to assess clinical severity in patients with BE. The clinical severity scoring system is made up of six items: wheezing, drawing, air intake, SaO2 (with and without O2 input), RR and HR. Each item is scored from 0 to 3, the values of each item are added and a total result of (0-5) mild, (6-10) moderate and (11-16) severe is obtained, with 16 being the maximum score and 0 the minimum. A higher clinical score indicates a worse condition.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Nicolas Mr Cuenca Zaldívar, Principal Investigator — Hospital Guadarrama, servicio de fisioterapia
Locations (1):
- J.Nicolas Cuenca Zaldivar, Guadarrama, Madrid, Spain

REFERENCES:
- [Derived] Roque-Figuls M, Gine-Garriga M, Granados Rugeles C, Perrotta C, Vilaro J. Chest physiotherapy for acute bronchiolitis in paediatric patients between 0 and 24 months old. Cochrane Database Syst Rev. 2023 Apr 3;4(4):CD004873. doi: 10.1002/14651858.CD004873.pub6. PMID 37010196